CLINICAL TRIAL: NCT01791010
Title: Respiratory Muscle Training in the Elderly: a Strategy for Preservation of Inspiratory and Expiratory Pressures Impacting on Mobility and Thickness of the Diaphragm.
Brief Title: Effects of Inspiratory Muscle Training in Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Helga Cecília Muniz de Souza, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IMT in elders
Record Dates: First submitted 2013-02-06; First posted 2013-02-13 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Muscular Atrophy; Sensitivity Training Groups; Aging
Keywords: Breathing exercises; Aged
MeSH Terms: conditions — Muscular Atrophy | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inspiratory muscle training (Experimental): Inspiratory muscle training for 8 weeks using a device that provides a linear resistance in the inspiratory phase. 7 days a week. 8 sets of 2 minutes twice a day. Intensity was at 40% of Maximal Inspiratory Pressure.
  Interventions: Other: Inspiratory muscle training
- Training sham (Sham Comparator): Training sham for 8 weeks using a device without provides resistance. 7 days a week. 8 sets of 2 minutes twice a day. Intensity was canceled.
  Interventions: Other: Training sham

INTERVENTIONS:
Other: Inspiratory muscle training
  Other Names: respiratory muscle training
  Arms: Inspiratory muscle training
Other: Training sham — Conducting fake training with the aim of blind the control group
  Arms: Training sham

SUMMARY:
Aging causes anatomical and physiological changes in the respiratory system and respiratory muscle strength with decline in its maximum function. This study aimed to evaluate the effects of inspiratory muscle training on respiratory muscle strength, thickness of the diaphragm and diaphragmatic mobility in older women. The investigators' hypothesis is that inspiratory muscle training improves respiratory muscle strength, the thickness of the diaphragm and diaphragmatic mobility in older women.

ELIGIBILITY:
Inclusion Criteria:

Elderly women are able to walk without aid and cognitive integrity.

Exclusion Criteria:

* Participation in other training or rehabilitation protocol;
* Contraindication or difficult to perform the evaluation;
* Difficulty adapting or adherence in training protocol;
* Smoking;
* Hemodynamic instability;
* Degenerative neuromuscular disease;
* Pulmonary comorbidities;
* Heart disease;
* Users of drugs that interfere in bone metabolism or muscle strength.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
respiratory muscle strength | Change from Baseline Respiratory Muscle Strength at 2 months

SECONDARY OUTCOMES:
Diafragmatic excursion and thickness of the diaphragm in the zone of apposition by ultrasonography | Change from Baseline Diafragmatic Excursion and Thickness of the Diaphragm at 2 months
  Ultrasound was used to evaluate diaphragm thickness non-invasively in the zone of apposition during tidal breathing and with changes in lung volume.
  During respiration to total lung capacity, measurement of the diafragmatic excursion was made by ultrasonography.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Background] Testa A, Soldati G, Giannuzzi R, Berardi S, Portale G, Gentiloni Silveri N. Ultrasound M-mode assessment of diaphragmatic kinetics by anterior transverse scanning in healthy subjects. Ultrasound Med Biol. 2011 Jan;37(1):44-52. doi: 10.1016/j.ultrasmedbio.2010.10.004. PMID 21144957
- [Background] Ueki J, De Bruin PF, Pride NB. In vivo assessment of diaphragm contraction by ultrasound in normal subjects. Thorax. 1995 Nov;50(11):1157-61. doi: 10.1136/thx.50.11.1157. PMID 8553271
- [Background] Enright SJ, Unnithan VB, Heward C, Withnall L, Davies DH. Effect of high-intensity inspiratory muscle training on lung volumes, diaphragm thickness, and exercise capacity in subjects who are healthy. Phys Ther. 2006 Mar;86(3):345-54. PMID 16506871